CLINICAL TRIAL: NCT05207319
Title: Effects of Integrated Moral Reasoning Development Intervention for Management of Violence in Schizophrenia: A Randomized Controlled Trial
Brief Title: Effects of Integrated Moral Reasoning Development Intervention for Management of Violence in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I-Shou University (Other)
Responsible Party: Principal Investigator, Mei-Chi Hsu, Professor, I-Shou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IShouU
Record Dates: First submitted 2021-12-27; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia; Moral Status; Violence
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the MRDI group (Moral Reasoning Development Intervention) (Experimental): The MRDI is comprised of 4 components that are run concurrently: moral reasoning, strategies of anger management and problem-solving and social skills.
  Interventions: Other: integrated Moral Reasoning Development Intervention (MRDI)
- the control group (No Intervention): The control group is the Treatment as Usual (TAU).

INTERVENTIONS:
Other: integrated Moral Reasoning Development Intervention (MRDI) — The MRDI is comprised of 4 components that are run concurrently: moral reasoning, strategies of anger management and problem-solving and social skills.
  Arms: the MRDI group (Moral Reasoning Development Intervention)

SUMMARY:
Moral cognition is an important and multidimensional, but often overlooked, determinant of violence. Very few interventions have systematically examined the role of moral reasoning, anger management and problem-solving together in violence. A randomized controlled trial was conducted to comprehensively evaluate the sustained effects of an integrated Moral Reasoning Development Intervention (MRDI) on management of repetitive violence in schizophrenia. This study placed special emphasis on essential components related to moral reasoning and violence in patients with schizophrenia. Evaluations including measures of violence, moral reasoning, ethical valuation and judgement, decision-making, conflict management style, and personality traits, were performed at baseline, end of intervention, and 1-month follow-up after intervention. MRDI was superior to treatment-as-usual in improving moral reasoning and related variables and violence outcomes. In comparison with the treatment-as-usual group, patients in the MRDI group showed improved levels of moral reasoning whereas decreased levels of violent behaviors. The MRDI participants also experienced significantly greater improvements or changes in their ethical valuation and judgement, decision-making style and preferences, and conflict management style. Our findings provide important implications for risk assessment and violence management and prevention.

DETAILED DESCRIPTION:
Moral cognition is an important and multidimensional, but often overlooked, determinant of violence. Very few interventions have systematically examined the role of moral reasoning, anger management and problem-solving together in violence. A randomized controlled trial was conducted to comprehensively evaluate the sustained effects of an integrated Moral Reasoning Development Intervention (MRDI) on management of repetitive violence in schizophrenia. This study placed special emphasis on essential components related to moral reasoning and violence in patients with schizophrenia. Evaluations including measures of violence, moral reasoning, ethical valuation and judgement, decision-making, conflict management style, and personality traits, were performed at baseline, end of intervention, and 1-month follow-up after intervention. MRDI was superior to treatment-as-usual in improving moral reasoning and related variables and violence outcomes (p < 0.05). In comparison with the treatment-as-usual group (n = 22), patients in the MRDI group (n = 21) showed improved levels of moral reasoning whereas decreased levels of violent behaviors. The MRDI participants also experienced significantly greater improvements or changes (p < 0.05) in their ethical valuation and judgement, decision-making style and preferences, and conflict management style. Our findings provide important implications for risk assessment and violence management and prevention.

The triggering point of violence is multi-faceted and dynamic. Many risk factors for violence intertwined and interacted at multiple levels. This integrated moral reasoning development intervention, when applied in conjunction with psychiatric standard care, could display synergistic and effective effects on moral reasoning and ethical evaluation, and impulsivity and personality features of repetitive violence in patients with schizophrenia. Suggestions for future research are made. There is a need to concurrently examine moral reasoning, violence and conflict handling styles in a dyadic context such as vSZ patients and their family members involved, so that a whole picture of the violence can be better observed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia for more than 2 years
* Psychiatrically hospitalized
* Repetitive violence within one year
* Having basic literacy
* More than 20 years old
* Less than 65 years old

Exclusion Criteria:

• Clinical diagnosis of catatonic schizophrenia and schizophreniform disorder.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The Adapted Version of the Sociomoral Reflection Measure | Change of status of moral reasoning from Baseline (T1), immediately after the intervention (T2), to 1-month follow-up after intervention (T3)
  Moral reasoning (The score 1 which corresponds with the first stage of Kohlberg's moral development, indicates the patient did not understand the moral content of the proposition. )
Multidimensional Ethics Scale | Change of ethical valuation from Baseline (T1), immediately after the intervention (T2), to 1-month follow-up after intervention (T3)
  Ethical valuation (The patients are required to rate the questionable actions of a hypothetical auditor on several 7-point Likert scales, anchored on such as unjust/just, unfair/fair, unethical/ethical, not morally right/morally right, culturally unacceptable/culturally acceptable.)
Rational Experiential Inventory | Change of reasoning and thinking styles from Baseline (T1), immediately after the intervention (T2), to 1-month follow-up after intervention (T3)
  Reasoning and thinking styles (A higher score indicates a more rational/experiential thinking style.)
Rahim Organizational Conflict Inventory-II | Change of conflict management style from Baseline (T1), immediately after the intervention (T2), to 1-month follow-up after intervention (T3)
  Conflict management style (The higher the score is, the greater a particular conflict management style is used.)
Modified Overt Aggression Scale | Aggression frequency at Baseline
  Aggression Frequency
Buss-Perry Aggression Questionnaire | Change of violence/aggression from Baseline (T1), immediately after the intervention (T2), to 1-month follow-up after intervention (T3)
  Violence/Aggression (The higher the score is, the higher the patient has the violent behavior.)
Ten Item Personality Inventory | Change of personality traits from Baseline (T1), immediately after the intervention (T2), to 1-month follow-up after intervention (T3)
  Personality traits (A greater change from the baseline in this scale (with higher score) on each of personality traits represents more the expression of each personality trait was calculated.)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chi Hsu, Ph.D, Principal Investigator — I-Shou University
Locations (1):
- I-Shou University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No